CLINICAL TRIAL: NCT04277741
Title: Long-term Consumption of Resistant Starch Type-4 (RS4): Implications for Obesity and Chronic Disease
Brief Title: Long-term Consumption of Resistant Starch Type-4 (RS4)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI departure from university
Sponsor: Kansas State University (Other)
Collaborators: MGP Ingredients, Inc. (Industry)
Responsible Party: Principal Investigator, Sara K Rosenkranz, Principal Investigator, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro9978
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Cholesterol, Elevated; Overweight or Obesity
MeSH Terms: conditions — Hypercholesterolemia; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will be blind to the condition that they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant starch bar (Experimental): The RS4 group will consume one nutrition bar per day formulated using Fibersym® RW.
  Interventions: Dietary Supplement: RS4 bar
- Native wheat bar (Active Comparator): The control group will consume one native wheat starch bar per day.
  Interventions: Dietary Supplement: Control bar

INTERVENTIONS:
Dietary Supplement: RS4 bar — The RS4 group will consume one nutrition bar per day formulated using Fibersym® RW containing 20g fiber.
  Arms: Resistant starch bar
Dietary Supplement: Control bar — The control group will consume one native wheat starch bar per day.
  Arms: Native wheat bar

SUMMARY:
The primary objective of the current proposal is to determine the effectiveness of long-term consumption of Fibersym® RW for improving blood lipids (including cholesterol) and body composition. The overall goal of this clinical research is to determine the potential effects that RS4 consumption may have on the prevention of obesity and obesity-related diseases. Fiber in the form of RS4 will be used for the proposed study, given that fiber has been shown to have many beneficial effects on modifiable risk factors associated with obesity-related diseases. Using a long-term randomized-controlled intervention design, blood lipids (total cholesterol, LDL-c, HDL-c, triglycerides) and body composition will be assessed. The investigators anticipate reductions in cholesterol and body fat percentage following 8-weeks of Fibersym® RW consumption.

DETAILED DESCRIPTION:
This study will investigate the metabolic effects of daily RS4 consumption in overweight and obese adults. The investigators will recruit approximately 50 (BMI: 23-34.9kg/m2) adults ages 18-65yrs, who have elevated to borderline-high LDL-cholesterol (116-159mg/dL) to an 8-week randomized controlled intervention. Participants will be recruited in three waves of 16 participants each. Following a 7-10-day run-in where fiber intake is monitored, participants will be randomized to either the control or the RS4 group. The RS4 group will consume a high fiber bar, daily, for 8-weeks that will contain approximately 60-70% of the daily reccomended allowance of fiber. The primary outcome for this study will be fasting plasma LDL-Cholesterol (LDL-c). Secondary outcomes include body composition following daily RS4 consumption for 8-weeks. All health assessments will be conducted before the intervention begins, at the 4-week mid-point, and immediately following the 8-week intervention. Participants will fast for 10 -12 hrs. before reporting to the PAN-CRC for each testing session. The meal consumed prior to each testing session will be standardized so that it does not vary within the individual between testing sessions.

Treatments. The two treatment conditions are RS4 and control. Participants will be asked to consume one nutrition bar as part of their breakfast each day with no other changes to their diet. The control group will consume one native wheat starch bar per day. The RS4 group will consume one nutrition bar per day formulated using Fibersym® RW containing 20g fiber. This amount would likely put individuals in the recommended dietary fiber intake range according to the dietary recommended intake ( Institutes of Medicine: 14g fiber/1000 kcal). All nutrition bars will contain the same ingredients and be matched for calories; however, fiber will vary between the bars.

Health assessments. The KSU Nutrition team will conduct all health assessments at each time point. Height (cm), weight (kg), and waist circumference (cm) will be measured to determine basic anthropometrics, and a dual-energy X-ray absorptiometry scan (DXA) will be used to determine body composition (body fat percentage and non-fat mass). Blood pressure (systolic and diastolic (mmHg) will be measured using a standard automated monitor. Fasting total cholesterol (TC), triglycerides (TRG), glucose, LDL-c, and HDL-c will be measured via an LDX Cholestech using a single venous blood draw for assessment. Plasma glucose and insulin will be determined via the same venous sample. Satiety will be measured during each testing session to determine how Fibersym® RW impacts feelings of fullness and hunger.

Compliance Checks. To ensure compliance with consumption of the nutrition bars provided, participants will be asked to return to the PAN-CRC to return any leftover bars at the end of each intervention week (if any remain), and to pick up a new supply of their assigned bar. Participants will also be given a checklist that indicates their daily consumption of the given bars. The checklist will include options such as: I consumed the 100% of the bar, forgot to consume, consumed part of the bar (with options to check a percent of the bar consumed). To ensure that habitual dietary intake is maintained, participants will be instructed to complete a 3-day dietary record (two weekdays and 1 weekend day) prior to each testing session, allowing the investigators to determine any dietary changes that may occur during the 8-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 23 kg/m2
* elevated to borderline-high LDL-cholesterol (116-159 mg/dL)

Exclusion Criteria:

* known allergy to wheat or gluten
* currently taking medication for chronic disease including anti-inflammatory, anti-hypertensive, lipid lowering, glucose controlling, or steroidal medications
* taking any supplements that may affect metabolism
* having anemia or a history of anemia
* current smoker or a user in the past three months
* currently pregnant or lactating/planning to become pregnant during the intervention
* having elevated blood pressure (≥130mmHg/≥80mmHg)
* presence of diagnosed diabetes mellitus, inflammatory disease, atherosclerotic disease, or other relevant chronic conditions that may affect metabolic processes
* total cholesterol ≥ 240mg/dL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in plasma lipids | Week 0, 4, and 8
  Total cholesterol (TC), LDL-c , VLDL-c, HDL-c , triglycerides (TG) from blood sample in a fasted state

SECONDARY OUTCOMES:
Change in body composition | Week 0, 4, and 8
  Percent body fat as measured by DXA scan
Change in BMI | Week 0, 4, and 8
  Weight and height will be combined to report BMI in kg/m^2
Change in homeostatic model assessment for insulin resistance (HOMA-IR) | Week 0,4, and 8
  Calculated from fasting glucose and insulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Sara Rosenkranz, PhD, Principal Investigator — Kansas State University
Locations (1):
- Physical Activity and Nutrition Clinical Research Consortium, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No